CLINICAL TRIAL: NCT01583010
Title: Improvement of Needle Visibility in In-line Regional Anaesthesia by "Advanced Needle Visualization Technology ®"
Brief Title: Improvement of Needle Visibility in Ultrasound Guided Regional Anaesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Hahn, Dr., Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EK572/2011
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Anaesthesia; Trauma
Keywords: ultrasound guided regional anaesthesia needle visualization
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment Group (No Intervention): Patients receiving ultrasound guided regional anaesthesia without using Advanced Needle Visualization Technology(R)
- ANV ® Group (Active Comparator): Patients receiving ultrasound guided regional anaesthesia with using Advanced Needle Visualization Technology(R)
  Interventions: Device: ANV(R)

INTERVENTIONS:
Device: ANV(R) — Device: Advanced Needle Visualization Technology ®
  Software update for SonoSites M-Turbo® and S-series™ ultrasound systems with enhanced 15-20Mhz ultrasound probe.
  Arms: ANV ® Group
  Other Names: SonoSite M-Turbo Mbe
  Arms: ANV ® Group

SUMMARY:
Needle tip visualization, although fundamental to the safety and efficacy of ultrasound-guided regional anesthesia (UGRA), can be extremely challenging. This problem is most marked at steep insertion angles. Studies in patients with UGRA demonstrate that echogenic needle designs have the potential to offer improved visibility and accuracy.

Our study pursues another approach. We use (for differentiation) echogenic nerve block needles with ANV®, a new SonoSite software-upgrade (Advanced Needle Visualization Technology®). We will compare UGRA with ANV® against standard UGRA without using this SonoSite software-upgrade. Patients undergoing femoral, supraclavicular or other nerve blocks as part of their routine anesthetic management are included.

This work represents the first randomized controlled double blinded clinical trial of ANV® in patients undergoing UGRA. We hypothesize, that we can decrease the time without needle visualization (Loss of needle time in percentage of procedure time) during in-line regional anaesthesia. Furthermore we will record quality of visibility, duration of procedure and insertion angle of the needle.

DETAILED DESCRIPTION:
Patients scheduled to undergo surgery with femoral (n = 50) and supraclavicular (n=50) anaesthesia (100 blocks total) gets included in this study. These 50 patients will be randomized equally using sealed opaque envelopes to two parallel groups: standard treatment UGRA (n=25) and SonoSites ANV® (n= 25) UGRA.

An experienced anaesthesiologist from department of anaesthesiology, general intensive care and pain medicine will perform UGRA. Because of safety reasons and best assessment of needle visibility all UGRA in this study are going to performed with in-plane ultrasound technique. Needle length and gauge are standardized.

The ultrasound imaging of each nerve block gets recorded onto a DVD for analysis. Recording of performed UGRA will start with placement of ultrasound probe and will finish with needle leaving the skin (procedure time), get stored, checked to exclude technical failures and analysed with a one second discrimination by two blinded observers for needle visibility. All information indicating ANV®-status on ultrasound image will be deleted. Hence for procedure and following analysis we will ensure that patient and the objective observer are blinded.

Images with full needle visibility will be related to images without needle visibility. Time of needle visibility will be described in percent of procedure time.

Enduring visualization of complete needle in ultrasound beam won't be given during the whole procedure. For differentiation of complete needle visibility, partial or no visibility in in-plane UGRA, we will use needles with ultrasound visible marks (echogenic needles). If the objective observers will visualize all 3 marks and pole of the needle in ultrasound-image, needle is completely in-plane and visible for analysis. For partial visibility of marks we will use a needle visibility grading dependent to number of visible marks (One mark = poor visibility, two marks = middle visibility, three marks=good visibility). If there won't be visible marks in ultrasound image, needle is in absence and gets evaluated as "not visible".

Dependent to position of anatomic target structure each nerve block will need a different angle of needle insertion. This measured angle will be used to compare times of needle visibility dependent to insertion angle of the needle. Significant differences may appear especially in steep angles of needle.

In this study we will use Naropin® (Ropivaciane, 7.5mg/ml) as local anaesthetic for all UGRA.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who give consent and undergo a femoral or supraclavicular nerve block.

Exclusion Criteria:

* Patients get excluded if they refused or are unable to give consent by other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Time of needle visibilty in ultrasound-image | At time of ultrasound guided regional anaesthesia
  Measure is given in percentage of procedure time

SECONDARY OUTCOMES:
Procedure time | At time of ultrasound guided regional anaesthesia
  Duration of placement of the ultrasound probe up to needle-removal out of the skin.
Angle of needle insertion | At time of ultrasound guided regional anaesthesia
  Measurement of puncture-angle between skin an needle in the ultrasound-image.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Hahn, Univ. Lektor Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Anesthesia, Intensive Care Medicine and Pain Therapy, Medical University Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Hebard S, Hocking G. Echogenic technology can improve needle visibility during ultrasound-guided regional anesthesia. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):185-9. doi: 10.1097/aap.0b013e31820d4349. PMID 21425515
- [Background] Maecken T, Zenz M, Grau T. Ultrasound characteristics of needles for regional anesthesia. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):440-7. doi: 10.1016/j.rapm.2007.07.002. PMID 17961844
- [Background] Chapman GA, Johnson D, Bodenham AR. Visualisation of needle position using ultrasonography. Anaesthesia. 2006 Feb;61(2):148-58. doi: 10.1111/j.1365-2044.2005.04475.x. PMID 16430568
- [Background] Chin KJ, Perlas A, Chan VW, Brull R. Needle visualization in ultrasound-guided regional anesthesia: challenges and solutions. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):532-44. doi: 10.1016/j.rapm.2008.06.002. PMID 19258968